CLINICAL TRIAL: NCT05302687
Title: Use of Probiotic to Modulate Vaginal Microflora and General Women's Health
Brief Title: Probiotic Modulates Vaginal Microflora
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Min-Tze LIONG (Other)
Collaborators: International Islamic University Malaysia (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IREC 2021-318
Record Dates: First submitted 2022-03-17; First posted 2022-03-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Microbial Colonization
Keywords: probiotics
MeSH Terms: conditions — Communicable Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A double-blind randomized placebo-controlled trial design has been chosen. Randomization for the parallel prevention phase will be carried out after checking the inclusion and exclusion criteria.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization will be performed by the study statistician, who had no contact with the participants. The allocation sequence will not available to any member of the research team until databases had been completed and locked. Since this is a double-blinded study, both the research team and subject will not know in which group the subject is assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic 9 log CFU/day (Experimental): Intervention consists of daily administration of one sachet/day of probiotic for 12 weeks, where each sachet contains 9 log CFU of probiotic.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): placebo contains primarily carrier and without probiotic. The placebo are identical in taste and appearance and appear as light-yellow powder.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — This project aims to evaluate differences in general women's health of women on probiotic and placebo via the use of questionnaire and evaluate differences in immunity of women on probiotic and placebo via blood immunity profiling. To evaluate differences in gut microbiota profiles of women on probiotic and placebo via blood fecal microbiota profiling.
  Arms: probiotic 9 log CFU/day
Dietary Supplement: placebo — This project aims to evaluate differences in general women's health of women on probiotic and placebo via the use of questionnaire and evaluate differences in immunity of women on probiotic and placebo via blood immunity profiling. To evaluate differences in gut microbiota profiles of women on probiotic and placebo via blood fecal microbiota profiling.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effects of oral administration of probiotic at 9 log colony forming unit (CFU)/day on vaginal microbiota profiles compared to placebo via the use of vaginal self-swab microbiota profiling.

DETAILED DESCRIPTION:
1. To evaluate differences in general women's health of women on probiotic and placebo via the use of questionnaire.
2. To evaluate differences in immunity of women on probiotic and placebo via blood immunity profiling.
3. To evaluate differences in gut microbiota profiles of women on probiotic and placebo via blood fecal microbiota profiling.

ELIGIBILITY:
Inclusion Criteria:

* Generally, healthy women aged 18-80. - Currently free from urogenital infections such as urinary tract infection (UTI), bacterial vaginosis (BV), or yeast vaginitis.
* Willing to commit throughout the experiment.

Exclusion Criteria:

* Pregnant.
* On vaginal suppository treatments within 4-weeks prior to entering the study.
* On oral medication for vaginal illnesses or any vaginal therapy such as hormones and estrogen within 4-weeks prior to entering the study.
* On long term medication (> 6 months) for any illnesses.
* Have used vaginal estrogen cream, ring or tablet within 4-weeks prior to entering the study.
* Have used vaginal moisturizers, lubricants or homeopathic preparations within 4-weeks prior to entering the study.
* Have used spermicide agent within 4-weeks prior to entering the study.
* Pelvic or any gynecologic surgery 6-months prior to entering the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
differences in general women's health | 12 weeks
  To evaluate differences in general women's health of women on probiotic and placebo via the use of the Women's Health Questionnaire (WHQ) questionnaire containing 37-items covering aspects of anxiety and depression, memory, sleep and sexual issues, on a 4-point Likert scale including some items with reverse scoring, with higher scores indicating poorer health status.
differences in immunity of women | 12 weeks
  To evaluate differences in immunity of women on probiotic and placebo in terms of blood immunity profiling via measuring concentrations of cytokines such as interleukin (IL)-1b using commercially available ELISA kit.
differences in gut microbiota profiles of women | 12 weeks
  To evaluate differences in gut microbiota profiles of women on probiotic and placebo via microbiota profiling using DNA of fecal samples amplified for bacterial 16S rRNA and analyzed for high-throughput community sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Syahril Azizan Azha, Doctor, Principal Investigator — IIUM Kuantan Campus
Locations (1):
- International Islamic University Malaysia, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nisaa AA, Mageswary U, Pei X, Kadir MN, Oon CE, Rajendran D, Tan JJ, Roslan FF, Balasubramaniam SD, Sany S, Ismail EHE, Azizan AS, Liong MT. Probiotic enhanced immunity and mental wellbeing of generally healthy women: a randomised, placebo-controlled and double-blind study. Benef Microbes. 2025 Feb 24;16(4):377-394. doi: 10.1163/18762891-bja00061. PMID 40008414